CLINICAL TRIAL: NCT03406897
Title: A Pilot, Safety and Feasibility Trial of High-Dose Omega-3 Fatty Acids and High-Dose Cholecalciferol (Vitamin D) Supplementation in Type 1 Diabetes
Brief Title: Pilot Study of OMEGA-3 and Vitamin D in High-Dose in Type I Diabetic Patients
Acronym: POSEIDON
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: Diabetes Research Institute Foundation (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180173
Record Dates: First submitted 2018-01-10; First posted 2018-01-23 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus; Diabetes, Autoimmune
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Diabetes Mellitus | interventions — Cholecalciferol; Vitamin D; Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: The study is a two-arm, open label, randomized trial. All four groups will receive standard intensive diabetes treatment with insulin and dietary management.
  Group I: Fourteen (14) adults (18-65 years) of established T1D > 6 months (>180 days) and up to 10 years of T1D duration Group II: Fourteen (14) adults (18-65 years) of new-onset T1D diagnosed within last 6 months (≤ 180 days) Group III: Fourteen (14) children (6-17 years) of established T1D > 6 months (>180 days) and up to 10 years of T1D duration Group IV: Fourteen (14) children (6-17 years) of new-onset T1D diagnosed within last 6 months (≤ 180 days)
  Participants in each group will be randomly assigned in a 1:1 ratio to receive either one year of high dose Omega-3 fatty acids and Vitamin D combination (Arm A) or Vitamin D alone (Arm B). Both arms will receive Vitamin D supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omega-3 and Vitamin D Combination (Active Comparator): The treatment arm A includes Omega-3 Fatty Acids and Cholecalciferol (Vitamin D) supplement.
  Interventions: Drug: Cholecalciferol; Drug: Omega 3 fatty acid
- Vitamin D Only (Active Comparator): The treatment arm B (control group) will receive only Cholecalciferol (Vitamin D) supplement.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Oral Administration
  Other Names: Vitamin D
Drug: Omega 3 fatty acid — Oral Administration
  Other Names: Omega 3
  Arms: Omega-3 and Vitamin D Combination

SUMMARY:
The investigator propose to test the safety and efficacy of a regimen that combines Omega-3 Fatty Acids and Vitamin D in a design that considers timing and duration of administration in relation to their effects and predicted synergies.

DETAILED DESCRIPTION:
These agents may afford promote sustained immune regulation, reduce inflammation, and provide support for the residual beta cell mass. This integrated therapeutic regimen addresses major pathogenic mechanisms in T1D (Type 1 Diabetes) and thus represents a rational and well supported approach to preserve insulin secretion in T1D (Type 1 Diabetes). This approach could halt the disease progress, preserve β-cell function and hopefully reduce dose of insulin required to manage T1D (Type 1 Diabetes). The investigator hypothesizes that Omega-3 Fatty Acids and Vitamin D, administered to patients with newly or established T1D (Type 1 Diabetes) and residual stimulated C-peptide secretion will be safe and may preserve insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible to participate in this study:

* Subject must be able to understand and provide informed consent.
* Males and females, 6-17 years for children and 18-65 years of age for adult group.
* For new onset T1D - from onset to 6 months (180 days) post-diagnosis at the time of randomization.
* For established T1D - At least 6 months and up to 10 years from the diagnosis at the time of randomization.
* Affected by T1D, according to ADA standard criteria, and confirmed by positivity of at least one T1D-associated autoantibody, to GAD65, IA-2, ZnT8, or insulin autoantibody (if patient has been treated with insulin for less than 2 weeks).
* T1D must be treated with insulin (except if participant is in Honeymoon period/phase).
* Stimulated C-peptide peak level, at the baseline 1 visit MMTT, ≥ 0.2 ng/ml.
* Female subjects of childbearing potential must have a negative pregnancy test upon study entry.
* Adequate venous access to support study required blood draws.

Exclusion Criteria:

Patients must not meet any of the following criteria to be eligible to participate:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
* BMI>30 kg/m2.
* Contra-indications to any of the drugs used in the trial (as per package insert, e.g., knowledge of hypersensitivity to drugs or its excipients).
* Uncompensated heart failure, fluid overload, myocardial infarction or liver disease or severe impairment of a vital organ within the last 6 weeks before enrollment.
* Any of the following laboratory findings indicating hemoglobin <10.0 g/dL; leukocytes <3,000/μL; neutrophils <1,500/μL; lymphocytes <800/μL; platelets <100,000/μL.
* Any sign or diagnosis of significant chronic active infection (e.g., hepatitis, tuberculosis, EBV, or CMV), or screening laboratory evidence consistent with a significant chronic active infection (such as positive for HIV, IGRA test for TB, or hepatitis B-C).
* Ongoing acute infections, e.g., acute respiratory tract, urinary tract, or gastrointestinal tract infections.
* Ongoing or anticipated use of diabetes medications other than insulin.
* Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within prior 7 days of screening.
* Recent recipient of any licensed or investigational live attenuated vaccine(s) within 6 weeks of randomization.
* Use of investigational drugs within 3 months of participation.
* Concomitant therapy with immunosuppressive drugs, immunomodulators, or cytotoxic agents, or previous therapy less than 3 months from randomization.
* History or diagnosis of malignancy, with the exception of a history of localized basal or squamous cell carcinoma.
* History of gastroparesis or other severe gastrointestinal disease..
* Presence of an allograft.
* AST, ALT or Alkaline Phosphatase >2 times upper limit of normal or total bilirubin >1.5 times upper limit of normal.
* History of mental illness deemed to be clinically unstable or any situation that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
* History of illicit drug or alcohol abuse.
* Pregnancy or ongoing breastfeeding for women; unwillingness or inability of both females and males of childbearing age to use a reliable and effective form of contraception, for the entire duration of the study.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camillo Ricordi, M.D., Study Director — Professor and Center Director of Diabetes Research Institute
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baidal DA, Ricordi C, Garcia-Contreras M, Sonnino A, Fabbri A. Combination high-dose omega-3 fatty acids and high-dose cholecalciferol in new onset type 1 diabetes: a potential role in preservation of beta-cell mass. Eur Rev Med Pharmacol Sci. 2016 Jul;20(15):3313-8. PMID 27467009

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
Started | 12 | 15
Completed | 7 | 8
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 12 | 22
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 6 | 7 | 13
  White, Hispanic | 5 | 7 | 12
  Asian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in MMTT (Mixed Meal Tolerance Test) 90 Min C-peptide
Description: Stimulated (90-minute sample of a MMTT) C-peptide at the 1-year visit greater or equal to baseline level measured by ng/mL.
  Change in 90-minute C-peptide between baseline and 1-year visit
Time Frame: Baseline and 1-Year Visit
Population: Group A: 7/12 subjects completed 1year follow-up. Group B: 8/15 subjects completed 1year follow up.
Measure: Median (Full Range); unit: ng/mL
Groups:
- Omega-3 and Vitamin D Combination: The treatment arm A includes Omega-3 Fatty Acids and Cholecalciferol (Vitamin D) supplement.
  Cholecalciferol: Oral Administration Omega 3 fatty acid: Oral Administration
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
Number analyzed (Participants) | 7 | 8
ng/mL | -1.23 [-1.60 to -0.17] | -0.62 [-1.44 to -0.15]

2. Secondary Outcome: Change in Hemoglobin A1c Level
Description: Change in HbA1c between baseline and 1-year
Time Frame: Baseline and 1-Year Visit
Population: Group A: 7/12 subjects completed 1year follow-up. Group B: 8/15 subjects completed 1year follow up.
Measure: Median (Full Range); unit: percentage of HbA1c
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
Number analyzed (Participants) | 7 | 8
percentage of HbA1c | 0.00 [-0.30 to 2.50] | -0.55 [-3.10 to 0.30]

3. Secondary Outcome: Change in Insulin Requirements
Description: Difference in insulin requirement at the 1-year visit compared to baseline measured in units/kg/day
Time Frame: Baseline and 1-Year Visit
Population: Group A: 7/12 subjects completed 1year follow-up. Group B: 8/15 subjects completed 1year follow up.
Measure: Median (Full Range); unit: units/kg/day
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
Number analyzed (Participants) | 7 | 8
units/kg/day | 0.16 [0.02 to 0.52] | 0.15 [-0.20 to 0.87]

4. Secondary Outcome: Number of Adverse Events (AE)
Description: Number of adverse events (AE) comparable to general diabetes population
Time Frame: Through study completion, and average of one year
Measure: Number; unit: number of adverse events
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
Number analyzed (Participants) | 12 | 15
number of adverse events | 31 | 28

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Omega-3 and Vitamin D Combination | Vitamin D Only
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/15
Other Adverse Events (participants affected / at risk) | 8/12 | 8/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 and Vitamin D Combination (N=12) | Vitamin D Only (N=15)
Acute perforated apendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetes Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 and Vitamin D Combination (N=12) | Vitamin D Only (N=15)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Right upper thigh abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Streptococcal pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
COVID-19 Infection (Infections and infestations) | 0 (0) | 3 (3)
Dyslipidemia (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 3 (19) | 3 (16) — Level 2 hypoglycemia
High Vitamin D levels (General disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperkalemia (General disorders) | 1 (1) | 0 (0)
Hyperphosphatemia (General disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oily rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza A (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Celiac Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated PT/INR (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Wisdom Teeth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03406897/Prot_SAP_000.pdf